CLINICAL TRIAL: NCT03499119
Title: A Phase I, Randomized, Open-label, Multiple-dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of AMG 334 in Children and Adolescents With Migraine
Brief Title: AMG 334 20160172 Pediatric Migraine PK Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20160172
Record Dates: First submitted 2018-03-07; First posted 2018-04-17 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Amelogenin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Other): Subjects with a body weight at Day 1 of less than weight threshold.
  Interventions: Drug: AMG 334 Dose 1; Drug: AMG 334 Dose 3
- Cohort 2 (Other): Subjects with a body weight at Day 1 of weight threshold or more.
  Interventions: Drug: AMG 334 Dose 1; Drug: AMG 334 Dose 2

INTERVENTIONS:
Drug: AMG 334 Dose 1 — Subjects weighing less than weight threshold at Day 1 will be randomized to either Dose 1 or Dose 3.
  Subjects weighing weight threshold or more at Day 1 will be randomized to either Dose 1 or Dose 2
Drug: AMG 334 Dose 2 — Subjects weighing weight threshold or more at Day 1 will be randomized to either Dose 1 or Dose 2.
  Arms: Cohort 2
Drug: AMG 334 Dose 3 — Subjects weighing less than weight threshold at Day 1 will be randomized to either Dose 1 or Dose 3.
  Arms: Cohort 1

SUMMARY:
AMG 334 20160172 Pediatric Migraine PK Study.

DETAILED DESCRIPTION:
An Open-label, Randomized, Multiple-dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of AMG 334 in Children and Adolescents With Migraine

ELIGIBILITY:
Inclusion Criteria:

* Subject's legally acceptable representative has provided informed consent and the subject has provided written assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated.
* Male and female children and adolescents ≥ 6 and <18 years of age upon entry into screening
* Diagnosis of migraines, with or without aura, according to the International Classification of Headache Disorders (ICHD 3rd Edition, 2013) for at least 12 months prior to the study screening
* Frequency of migraine of ≥ 4 migraine days per month in each of the 3 months prior to the study screening period

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study
* History of migraine with brainstem aura or hemiplegic migraine headache
* Medical history or other condition that compromises the ability of the subject or legally acceptable representative to give appropriate informed consent and/or assent
* Malignancy except non-melanoma skin cancers or cervical cancer in situ within the last 5 years.
* Presence of any clinical condition that in opinion of the investigator might increased the risk of subjects participating in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (14):
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - CarePoint, Englewood, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Synergy Health, Bradenton, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - PANDA Neurology and Atlanta Headache Specialists, Atlanta, Georgia
  - Riley Hosptial, Indianapolis, Indiana
  - Clinical Research Institute Inc, Plymouth, Minnesota
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Meridian Clinical Research, Hastings, Nebraska
  - Dent Neurosciences Research Center, Amherst, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Hershey AD, Paiva da Silva Lima G, Pannacciulli N, Mackowski M, Koukakis R, McVige JW. Pharmacokinetics and safety of erenumab in pediatric patients with migraine: A phase I, randomized, open-label, multiple-dose study. Clin Transl Sci. 2024 Mar;17(3):e13755. doi: 10.1111/cts.13755. PMID 38476099
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 63 participants screened, 53 participants were enrolled at 9 centers in the United States between 04 May 2018 and 23 November 2021. Enrollment was staggered by age category with adolescents 12 to < 18 years of age starting enrollment first, followed by children 6 to < 12 years of age.
Pre-assignment Details: Participants weighing < 40 kg (Cohort 1) received a dose of either 35 mg or 70 mg erenumab. Participants weighing ≥ 40 kg (Cohort 2) received a dose of either 70 mg or 140 mg erenumab. All participants participated in the initial treatment phase for a total of 12 weeks of treatment. Adolescents 12 to < 18 years of age at time of consent had the option of continuing treatment with the same dose they received in the initial treatment phase in a 40-week extension phase.
Groups:
- Cohort 1: Erenumab 35 mg: Participants weighing < 40 kg received a dose of 35 mg erenumab Q4W via SC injection in the initial 12-week treatment phase.
  Adolescents 12 to < 18 years of age at time of consent had the option of continuing treatment with the same dose they received in the initial treatment phase in a 40-week extension phase, for a total of 52 weeks of treatment.
- Cohort 1: Erenumab 70 mg: Participants weighing < 40 kg received a dose of 70 mg erenumab Q4W via SC injection in the initial 12-week treatment phase.
  Adolescents 12 to < 18 years of age at time of consent had the option of continuing treatment with the same dose they received in the initial treatment phase in a 40-week extension phase, for a total of 52 weeks of treatment.
- Cohort 2: Erenumab 70 mg: Participants weighing ≥ 40 kg received a dose of 70 mg erenumab Q4W via SC injection in the initial 12-week treatment phase.
  Adolescents 12 to < 18 years of age at time of consent had the option of continuing treatment with the same dose they received in the initial treatment phase in a 40-week extension phase, for a total of 52 weeks of treatment.
- Cohort 2: Erenumab 140 mg: Participants weighing ≥ 40 kg received a dose of 140 mg erenumab Q4W via SC injection in the initial 12-week treatment phase.
  Adolescents 12 to < 18 years of age at time of consent had the option of continuing treatment with the same dose they received in the initial treatment phase in a 40-week extension phase, for a total of 52 weeks of treatment.
Period: Initial Treatment Phase
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Started | 4 | 9 | 8 | 32
Completed | 3 | 9 | 7 | 29
Not Completed | 1 | 0 | 1 | 3
Not completed — Protocol Specified Criteria | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Decision by Sponsor | 1 | 0 | 1 | 1
Period: Optional Extension Phase
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Started (Enrollment into the extension phase was optional.) | 1 | 3 (One participant (6 to < 12 years of age) incorrectly received investigational product in the Optional Extension Phase.) | 5 | 27
Completed | 1 | 2 | 5 | 21
Not Completed | 0 | 1 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5
Not completed — Protocol Specified Criteria | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg | Total
Number analyzed (Participants) | 4 | 9 | 8 | 32 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (1.7) | 10.4 (1.0) | 14.6 (1.3) | 15.4 (1.5) | 14.1 (2.5)
Age, Customized [Count of Participants; unit: Participants]
  Children (6 to < 12 years) | 3 | 7 | 0 | 0 | 10
  Adolescents (12 to < 18 years) | 1 | 2 | 8 | 32 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 23 | 31
  Male | 3 | 6 | 4 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 4
  Not Hispanic or Latino | 3 | 8 | 8 | 30 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black (or African American) | 0 | 2 | 1 | 4 | 7
  Multiple | 0 | 0 | 0 | 2 | 2
  White | 4 | 6 | 7 | 26 | 43
  Other | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Maximum Concentration (Tmax) of Erenumab
Description: Blood samples for pharmacokinetic (PK) testing were collected for the measurement of PK concentrations. Serum erenumab concentrations were determined using a validated assay. Noncompartmental analysis (NCA) was performed for erenumab PK parameter estimation.
Time Frame: First dose: Days 1 (pre-dose), 8, 15, and 29 (pre-dose); third dose: Days 57 (pre-dose), 64, 71, and 85
Population: The PK analysis set contained all randomized participants who received at least 1 dose of erenumab and had at least 1 PK concentration result. Data were excluded from the NCA if:
  * participants missed the previous dose or the actual time deviated by > 30% from the nominal sample collection time
  * PK profile was missing > 2 samples
  * PK values at the beginning or end of PK profile were missing, or
  * predose PK sample concentration was > 5% of maximum concentration value.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 3 | 9 | 8 | 30
days
  First Dose | 7.0 [2.9 to 7.2] | 7.0 [2.9 to 14.0] | 9.0 [2.9 to 15.0] | 7.0 [2.9 to 16.0]
  Third Dose: number analyzed (Participants) | 3 | 9 | 7 | 27
  Third Dose | 7.2 [7.0 to 8.0] | 10.0 [7.0 to 21.0] | 9.0 [6.0 to 26.0] | 7.2 [4.0 to 15.0]

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Erenumab
Description: Blood samples for PK testing were collected for the measurement of PK concentrations. Serum erenumab concentrations were determined using a validated assay. NCA was performed for erenumab PK parameter estimation.
Time Frame: First dose: Days 1 (pre-dose), 8, 15, and 29 (pre-dose); third dose: Days 57 (pre-dose), 64, 71, and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 3 | 9 | 8 | 30
μg/mL
  First Dose | 7.92 (0.947) | 13.3 (4.85) | 7.16 (1.76) | 13.4 (4.53)
  Third Dose: number analyzed (Participants) | 3 | 9 | 7 | 27
  Third Dose | 11.3 (3.14) | 18.9 (7.29) | 14.1 (5.54) | 23.7 (8.83)

3. Primary Outcome: Trough Concentration (Ctrough) of Erenumab
Description: as for outcome 2
Time Frame: First dose: Days 1 (pre-dose), 8, 15, and 29 (pre-dose); third dose: Days 57 (pre-dose), 64, 71, and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 3 | 9 | 8 | 31
μg/mL
  First Dose | 3.92 (0.626) | 7.02 (2.85) | 4.23 (1.05) | 7.77 (2.79)
  Third Dose: number analyzed (Participants) | 3 | 9 | 7 | 29
  Third Dose | 5.43 (0.861) | 10.3 (5.47) | 9.81 (2.37) | 14.9 (5.87)

4. Primary Outcome: Area Under the Concentration Time Curve From 0 to 28 Days (AUC0-28day) of Erenumab
Description: as for outcome 2
Time Frame: First dose: Days 1 (pre-dose), 8, 15, and 29 (pre-dose); third dose: Days 57 (pre-dose), 64, 71, and 85
Population: as for outcome 1
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 3 | 6 | 6 | 21
day*μg/mL
  First Dose: number analyzed (Participants) | 2 | 6 | 6 | 19
  First Dose | 175 [165 to 185] | 282 [65.8 to 357] | 151 [112 to 192] | 277 [175 to 551]
  Third Dose: number analyzed (Participants) | 3 | 6 | 5 | 21
  Third Dose | 243 [176 to 269] | 465 [336 to 667] | 329 [180 to 437] | 475 [259 to 1000]

5. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant. A TEAE was defined as an AE starting on or after first dose of investigational product. The event did not necessarily have a causal relationship with study treatment.
Time Frame: Up to Week 52 + 16-week safety follow-up
Population: The safety analysis set consisted of all randomized participants who received at least 1 dose of erenumab during the initial treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 4 | 9 | 8 | 32
Participants | 2 | 6 | 6 | 28

6. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Measurements
Description: The following measurements were performed: systolic/diastolic blood pressure, heart rate, and temperature.
Time Frame: Up to Week 52 + 16-week safety follow-up
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 4 | 9 | 8 | 32
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Measurements
Description: Clinically significant changes in ECG was defined as incidence of abnormal ECG diagnosis based on 12-lead ECG including heart rate, QRS, QTc and PR intervals.
Time Frame: Up to Week 52
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 4 | 9 | 8 | 32
Participants | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Safety Tests
Description: The clinical laboratory safety tests included: chemistry, hematology, and urinalysis.
Time Frame: Up to Week 52 + 16-week safety follow-up
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 4 | 9 | 8 | 32
Participants | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Changes in Neurological Assessments
Description: The neurological examinations were completed as per standard of care.
Time Frame: Up to Week 52 + 16-week safety follow-up
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Erenumab 35 mg | Cohort 1: Erenumab 70 mg | Cohort 2: Erenumab 70 mg | Cohort 2: Erenumab 140 mg
Number analyzed (Participants) | 4 | 9 | 8 | 32
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Initial treatment phase: up to Week 12 + 16-week safety follow-up; optional extension phase: Week 12 to Week 52 + 16-week safety follow-up
Description: The safety analysis set consisted of all randomized participants who received at least 1 dose of erenumab during the initial treatment phase.
Groups:
- Initial Treatment Phase Cohort 1: Erenumab 35 mg: Participants weighing < 40 kg received a dose of 35 mg erenumab Q4W via SC injection in the initial 12-week treatment phase.
- Initial Treatment Phase Cohort 1: Erenumab 70 mg: Participants weighing < 40 kg received a dose of 70 mg erenumab Q4W via SC injection in the initial 12-week treatment phase.
- Initial Treatment Phase Cohort 2: Erenumab 70 mg: Participants weighing ≥ 40 kg received a dose of 70 mg erenumab Q4W via SC injection in the initial 12-week treatment phase.
- Initial Treatment Phase Cohort 2: Erenumab 140 mg: Participants weighing ≥ 40 kg received a dose of 140 mg erenumab Q4W via SC injection in the initial 12-week treatment phase.
- Optional Extension Phase Cohort 1: Erenumab 35 mg: Adolescents 12 to < 18 years of age at time of consent weighing < 40 kg continued to receive a dose of 35 mg erenumab Q4W via SC injection in the 40-week extension phase.
- Optional Extension Phase Cohort 1: Erenumab 70 mg: Adolescents 12 to < 18 years of age at time of consent weighing < 40 kg continued to receive a dose of 70 mg erenumab Q4W via SC injection in the 40-week extension phase.
- Optional Extension Phase Cohort 2: Erenumab 70 mg: Adolescents 12 to < 18 years of age at time of consent weighing ≥ 40 kg continued to receive a dose of 70 mg erenumab Q4W via SC injection in the 40-week extension phase.
- Optional Extension Phase Cohort 2: Erenumab 140 mg: Adolescents 12 to < 18 years of age at time of consent weighing ≥ 40 kg continued to receive a dose of 140 mg erenumab Q4W via SC injection in the 40-week extension phase.
Arm/Group | Initial Treatment Phase Cohort 1: Erenumab 35 mg | Initial Treatment Phase Cohort 1: Erenumab 70 mg | Initial Treatment Phase Cohort 2: Erenumab 70 mg | Initial Treatment Phase Cohort 2: Erenumab 140 mg | Optional Extension Phase Cohort 1: Erenumab 35 mg | Optional Extension Phase Cohort 1: Erenumab 70 mg | Optional Extension Phase Cohort 2: Erenumab 70 mg | Optional Extension Phase Cohort 2: Erenumab 140 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9 | 0/8 | 0/32 | 0/1 | 0/3 | 0/5 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9 | 1/8 | 1/32 | 0/1 | 1/3 | 0/5 | 1/27
Other Adverse Events (participants affected / at risk) | 2/4 | 6/9 | 6/8 | 19/32 | 0/1 | 2/3 | 4/5 | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Phase Cohort 1: Erenumab 35 mg (N=4) | Initial Treatment Phase Cohort 1: Erenumab 70 mg (N=9) | Initial Treatment Phase Cohort 2: Erenumab 70 mg (N=8) | Initial Treatment Phase Cohort 2: Erenumab 140 mg (N=32) | Optional Extension Phase Cohort 1: Erenumab 35 mg (N=1) | Optional Extension Phase Cohort 1: Erenumab 70 mg (N=3) | Optional Extension Phase Cohort 2: Erenumab 70 mg (N=5) | Optional Extension Phase Cohort 2: Erenumab 140 mg (N=27)
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Phase Cohort 1: Erenumab 35 mg (N=4) | Initial Treatment Phase Cohort 1: Erenumab 70 mg (N=9) | Initial Treatment Phase Cohort 2: Erenumab 70 mg (N=8) | Initial Treatment Phase Cohort 2: Erenumab 140 mg (N=32) | Optional Extension Phase Cohort 1: Erenumab 35 mg (N=1) | Optional Extension Phase Cohort 1: Erenumab 70 mg (N=3) | Optional Extension Phase Cohort 2: Erenumab 70 mg (N=5) | Optional Extension Phase Cohort 2: Erenumab 140 mg (N=27)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 4
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site warmth (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 7
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
QRS axis abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 1 | 1 | 6 | 0 | 0 | 1 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03499119/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT03499119/SAP_001.pdf